CLINICAL TRIAL: NCT06087263
Title: Phase 2 Study to Evaluate the Efficacy of Regorafenib in Specific GIST Mutation Subsets (KIT Exon 17, 18, or 14 Mutation and SDHB Deficient GIST) in the Post-imatinib Second-line Setting.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0390; NCI-2023-08857 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-10-12; First posted 2023-10-17 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Regorafenib (Experimental)
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — Given by PO
  Other Names: Stivarga®

SUMMARY:
To learn if regorafenib can help to control the disease.

DETAILED DESCRIPTION:
Primary Objectives:

To assess efficacy of regorafenib in second-line GIST for patients with KIT exon 17, 18, or 14 mutation and SDHB deficient who progressed on imatinib as measured by PFS (RECIST 1.1).

Secondary Objectives:

1. RR by RECIST 1.1 and CHOI criteria
2. Progression-free rate at 1 year and 2 years
3. Median OS and OS at 1 years, 2years, and 5 years

Exploratory objectives:

1. Resistance mechanism (ctDNA analysis) in patients initially responding to regorafenib
2. Response data on next line of treatment post regorafenib

ELIGIBILITY:
Inclusion Criteria:

Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for nonnodal lesions and short axis for nodal lesions) as≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam.

* Age ≥18 years.
* Histologic diagnosis of GIST with presence of KIT exon 17, 18, or 14 mutation, or SDHB deficiency on tumor biopsy and/ or liquid biopsy.
* Participants must have unresectable or metastatic GIST and radiologic progression on imatinib treatment. Imatinib treatment must have been discontinued at least 5 days prior to the first dose of study drug. All imatinib treatment will be counted as 1 line of therapy.
* ECOG performance status ≤2 (Karnofsky ≥60%) at screening.
* Life expectancy of at least 12 weeks (3 months).
* Subjects must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trialspecific procedure.
* Patients must have adequate organ and marrow function as definedbelow:

Hemoglobin ≥8 g/dL Absolute neutrophil count ≥1,000/mcL Platelets ≥100,000/mcL Total bilirubin ≤2 x institutional upper limit of normal (ULN) or <3 x ULN in the presence of Gilbert's Disease AST and ALT ≤3 × institutional ULN ALT and AST ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer) Alkaline phosphatase ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer) Serum creatinine ≤ 3 x the ULN or 24-hr creatinine clearance >30 ml/min (Cockcroft formula) INR/ PTT ≤ 1.5 x ULN. (Subjects who are prophylactically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care

* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women (defined as no menses for at least

  1 year) and surgically sterilized women are not required to undergo a pregnancy test.
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 2 months after the last dose of study drug.

Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately

• Subject must be able to swallow and retain oral medication.

Exclusion Criteria:

* Patients who had received treatment with TKI other than imatinib
* Uncontrolled hypertension (systolic pressure >140 mm Hg or diastolic pressure > 90 mm Hg [NCI-CTCAE v4.0] on repeated measurement) despite optimal medical management.
* Active or clinically significant cardiac disease including:

  * Congestive heart failure - New York Heart Association (NYHA) > Class II.
  * Active coronary artery disease.
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin.
  * Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before randomization, or myocardial infarction within 6 months before randomization.
* Evidence or history of bleeding diathesis or coagulopathy.
* Any hemorrhage or bleeding event ≥ NCI CTCAE v 5.0 Grade 3 within 4 weeks prior to start of study medication.
* Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism within 6 months of informed consent.
* Patients with any previously untreated or concurrent cancer that is distinct in primary site or histology except cervical cancer in-situ, treated ductal carcinoma in situ of the breast, curatively treated nonmelanoma skin carcinoma, noninvasive aerodigestive neoplasms, or superficial bladder tumor. Subjects surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before registration are allowed. All cancer treatments must be completed at least 3 years prior to registration.
* Patients with pheochromocytoma.
* Patients with evidence of chronic hepatitis B virus (HBV) infection (except HBV viral load is undetectable on suppressive therapy)
* Patients with a history of hepatitis C virus (HCV) infection (Except the patients have been treated and cured or are currently on treatment with an undetectable HCV viral load)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Ongoing infection > Grade 2 NCI-CTCAE v5.0.
* Symptomatic metastatic brain or meningeal tumors.
* Presence of a non-healing wound, non-healing ulcer, or bone fracture.
* Major surgical procedure or significant traumatic injury within 28 days before start of study medication (minor surgical procedures such as central venous catheter placement, tumour needle biopsy, and feeding tube placement are not considered major surgical procedures).
* Renal failure requiring hemo-or peritoneal dialysis.
* Dehydration Grade >1 NCI-CTCAE v5.0.
* Patients with seizure disorder requiring medication.
* Persistent proteinuria Grade 3 NCI-CTCAE v5.0 (> 3.5 g/24 hrs, measured by urine protein: creatinine ratio on a random urine sample).
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
* Pleural effusion or ascites that causes respiratory compromise (≥ NCI-CTCAE version 5.0 Grade 2 dyspnea).
* History of organ allograft (including corneal transplant).
* Any malabsorption condition.
* Women who are pregnant or breast-feeding.
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
* Pregnant women, as documented by a serum beta human chorionic gonadotropin (β-hCG) pregnancy test obtained within 7 days before treatment consistent with pregnancy, are excluded from this study because regorafenib has evidence of the potential for teratogenic or abortifacient effects in animal studies. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with regorafenib, breastfeeding should be discontinued if the mother is treated with regorafenib. Females of non-childbearing potential (postmenopausal for more than 1 year; bilateral tubal ligation; bilateral oophorectomy; hysterectomy) do not require a serum β-hCG test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2032-07-01 (Estimated); Study Completion 2034-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Neeta Somaiah, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org